CLINICAL TRIAL: NCT01272310
Title: A Phase I/II, Open Clinical Trial to Assess the Safety, Tolerability and Efficacy of a Fixed Dose Combination Therapy of: Hydroxychloroquine (HCQ), Pegylated Interferon Alpha-2a (Peg-IFN Alpha-2a) and Ribavirin (RBV) in Chronic Hepatitis C Genotype 1 Infected Subjects Who Failed to Respond Following a Course of Peg-IFN and RBV Therapy (SoC).
Brief Title: Clinical Trial to Assess Safety and Efficacy of Combination Therapy: Hydroxychloroquine, Pegylated Interferon Alpha-2a and Ribavirin in Chronic Hepatitis C Subjects Non-responders to the Standard of Care Therapy.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Dr. Yaakov Maor, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-10-8033-YM-CTIL; HCQ-001-IL
Record Dates: First submitted 2011-01-03; First posted 2011-01-07 (Estimated); Last update posted 2011-01-07 (Estimated); Status verified 2011-01

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic Hepatitis C; Combination Therapy; Hydroxychloroquine; Pegylated Interferon Alpha-2a; Ribavirin; Chronic Hepatitis C Genotype 1 infected adult subjects
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Hydroxychloroquine; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Combination therapy (Experimental)
  Interventions: Biological: Hydroxychloroquine (HCQ), Pegylated Interferon Alpha-2a (Peg-IFN alpha-2a) and Ribavirin

INTERVENTIONS:
Biological: Hydroxychloroquine (HCQ), Pegylated Interferon Alpha-2a (Peg-IFN alpha-2a) and Ribavirin — HCQ will be taken daily as an oral tablet of 200 mg b.i.d. Pegylated Interferon Alpha-2a - (180 µg) will be administered as weekly subcutaneous (s.c.) injections of 0.5 ml.
  Ribavirin - will be taken daily based on the patient body weight. If body weight is < 75 kg, the total daily dose of Copegus® is 1000 mg, administered as 400 mg (2 tablets of 200 mg, morning intake) and 600 mg (3 tablets of 200 mg, evening intake). If body weight is >= 75 kg, the total daily dose is 1200 mg administered as twice 600 mg (3 tablets of 200 mg per intake, morning and evening).
  Other Names: Copegus; Pegasys

SUMMARY:
The study is aimed to investigate the safety, tolerability and efficacy of a fixed dose combination therapy of: Hydroxychloroquine (HCQ), Pegylated Interferon Alpha-2a (PEG-IFN alpha-2a) and Ribavirin (RBV) in Chronic Hepatitis C Genotype 1 Infected adult subjects who failed to respond following a course of PEG-IFN and RBV Therapy.

DETAILED DESCRIPTION:
This is a phase I/II, open clinical trial to assess the safety, tolerability and preliminary efficacy data of a fixed dose combination therapy of: HCQ, Peg-IFN alpha-2a and RBV in chronic hepatitis C genotype 1 infected subjects who failed to respond following a course of Peg-IFN and RBV Therapy (SoC). The study is a single center trial to be conducted at the Department of Gastroenterology & Hepatology, at Sheba Medical Center, Tel Hashomer, Israel.

Overall, thirty six (36) patients will be recruited. All patients enrolled will have a documented history of chronic HCV disease and being non-responder on earlier Peg-IFN based treatment lasting for at least 12 consecutive weeks prior to study enrolment.

The expected duration of patient screening period prior to enrollment into this study is in-between six weeks (42 days) up to 2 days prior to the study enrollment day at visit 2 (verification of compliance with inclusion/exclusion criteria including clinical laboratory results). Eligible patients will be enrolled into the study and will be observed twice on the first week of the study, once a week during the initiation of the treatment period at weeks 2,3 and week 4, later during the treatment period once a month at weeks 8-48 and at two follow up visits post treatment to take place at week 60 and 72 (allowing a time window of ± 5 days for all visits).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 18 and 70 years old.
2. Subjects diagnosed to have positive HCV antibodies using a third generation test.
3. Subject is diagnosed to have detectable HCV RNA by PCR.
4. Liver biopsy or FibroTest showing a METAVIR score ≥F2 and/or ≥A2.
5. Subject diagnosed to have compensated liver disease.
6. Subject is non-responder (null or partial) on prior Peg-IFN and RBV based treatment lasting for at least 12 consecutive weeks.
7. Treatment not discontinued due to intolerability to Peg-IFN or RBV.
8. Subjects able to comprehend and give informed consent for participation in this study.
9. Subject is willing to be treated and commit to all visits.

Exclusion Criteria:

1. Anti HCV therapy contraindications.
2. Subject is identified as a relapser on prior Peg-IFN and RBV based treatment.
3. Hypersensitivity to one of the three drugs (HCQ, Peg-IFN, RBV).
4. Patient has Anaemia,neutropenia, thrombocytopenia, elevated bilirubin levels, elevated ALT and/or AST, or elevated creatinin and INR greater than 1.5.
5. Concomitant liver disease other than hepatitis C: chronic hepatitis B, alcoholic liver disease, autoimmune hepatitis, Wilson's disease, hemochromatosis, alpha-1 antitrypsin deficiency.
6. Decompensated cirrhosis (Child Pugh >A).
7. Clinical evidence for hepatocellular carcinoma.
8. Human immunodeficiency virus co-infection.
9. Major uncontrolled psychiatric illness. Minor or situational depressions are allowed.
10. Active elicit drug or alcohol abuse.
11. Serious co-morbid conditions as: heart failure, significant coronary heart disease, chronic obstructive pulmonary disease, renal insufficiency, poorly controlled diabetes, autoimmune disorders, and malignant diseases in the previous 5 years.
12. Immunosuppressive treatment including corticosteroids,
13. Untreated or uncontrolled or thyroid disease.
14. Solid transplant organ (renal, heart, or lung).
15. Pregnancy or unwillingness to practice double contraception or abstinence by the subject of childbearing potential or partner.
16. Subject objects to the study protocol.
17. Concurrent participation in any other clinical study within 30 days prior to enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-01 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in physical examination | Twice on study first week , once a week during treatment initiation at weeks 2,3 ,4, later during treatment period once a month at weeks 8-48 and at weeks 60 and 72 follow up visits post treatment
  Body system screaning
Change from baseline in vital Signs | Twice on study first week , once a week during treatment initiation at weeks 2,3 ,4, later during treatment period once a month at weeks 8-48 and at weeks 60 and 72 follow up visits post treatment
  Heart Rate, Blood Presure, Respiratory Rate , Body temperature
Change from baseline in clinical laboratory parameters | Twice on study first week , once a week during treatment initiation at weeks 2,3 ,4, later during treatment period once a month at weeks 8-48 and at weeks 60 and 72 follow up visits post treatment
  Hematology, Blood Chemistry, Coagulation parameters, Urinalysis
Change from baseline in adverse events | Twice on study first week , once a week during treatment initiation at weeks 2,3 ,4, later during treatment period once a month at weeks 8-48 and at weeks 60 and 72 follow up visits post treatment
  All observed and or reported adverse events

SECONDARY OUTCOMES:
HCV RNA level | at 4,12, 24, 48 and 72 weeks after treatment
  Changes in HCV RNA levels, monitored along the study period. The efficacy of a HCQ-containing treatment regimen defined as the proportion of subjects with SVR i.e. undetectable HCV RNA <50 IU/ml) at 5 different time points: cEVR at 12 weeks, 4 weeks, 24 weeks, 48 weeks after treatment initiation and at 24 weeks after end of treatment (week 72).